CLINICAL TRIAL: NCT03417661
Title: An Evaluation of the Efficacy of HEXI-PREP by Clinell Wipes Versus Placebo and Chloraprep, for Use in Preoperative Skin Preparation
Brief Title: An Evaluation of the Efficacy of HEXI-PREP by Clinell Wipes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gama Healthcare Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GH001
Record Dates: First submitted 2018-01-09; First posted 2018-01-31 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Antimicrobial Effect

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HEXI-PREP By Clinell Wipes vs Placebo (Experimental): Both trial products will be applied bilaterally to between one and four predetermined anatomical sites on each participant, depending on whether the inclusion criteria for bioburden has been met for each sampling site. Each site will be sampled for bacterial load at four predetermined time points.
  Interventions: Drug: HEXI-PREP By Clinell Wipes; Drug: Placebos
- HEXI-PREP By Clinell Wipes vs Chloraprep (Experimental): Both trial products will be applied bilaterally to between one and four predetermined anatomical sites on each participant, depending on whether the inclusion criteria for bioburden has been met for each sampling site. Each site will be sampled for bacterial load at four predetermined time points.
  Interventions: Drug: HEXI-PREP By Clinell Wipes; Drug: Chloraprep
- Chloraprep vs Placebo (Experimental): Both trial products will be applied bilaterally to between one and four predetermined anatomical sites on each participant, depending on whether the inclusion criteria for bioburden has been met for each sampling site. Each site will be sampled for bacterial load at four predetermined time points.
  Interventions: Drug: Chloraprep; Drug: Placebos

INTERVENTIONS:
Drug: HEXI-PREP By Clinell Wipes — Sterile single sachet wipe containing 3ml solution.
  Arms: HEXI-PREP By Clinell Wipes vs Chloraprep; HEXI-PREP By Clinell Wipes vs Placebo
Drug: Chloraprep — Sterile applicator containing 3ml solution.
  Arms: Chloraprep vs Placebo; HEXI-PREP By Clinell Wipes vs Chloraprep
Drug: Placebos — Sterile saline (0.9% w/v) wipe, containing 3ml of solution.
  Arms: Chloraprep vs Placebo; HEXI-PREP By Clinell Wipes vs Placebo

SUMMARY:
This study evaluates the antimicrobial properties of HEXI-PREP by Clinell compared to both a negative and a positive control product.

DETAILED DESCRIPTION:
HEXI-PREP by Clinell is a sterile single sachet wipe containing chlorhexidine gluconate and isopropyl alcohol. Both active ingredients are well-established ingredients commonly used for their disinfectant properties.

This trial is designed to assess the superiority of HEXI-PREP by Clinell Wipe against a negative control, and also to demonstrate the relative efficacy of HEXI-PREP by Clinell WIpe against a similar commercially available product.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 - 70 years, who have provided written informed consent to participate in the study
* Test sites with a bacterial baseline count of ≥ 5.0 log10/cm2 at the inguinal (groin) test administration sites. ≥4.0 log10/cm2 at the abdominal test site and >3.0 log10/cm2 at the clavicular and/or median cubital regions at Day - 5 of screening
* Participants, who in the opinion of the Investigator, are in suitable health for inclusion in the study.

Exclusion Criteria:

* Exposure of the test sites to strong detergents, solvents or other irritants during the 14- day pre-test conditioning period or during the test period.
* Use of systemic or topical antibiotic medications, steroid medications or any other product known to affect the normal microbial flora of the skin, up to 1 month prior to the screening period, during the 14-day pre-test conditioning period or during the test period.
* Any known allergies to latex (rubber), alcohols, tape adhesives or to common antibacterial agents found in soaps, lotions or ointments, particularly chlorhexidine gluconate or chlorine.
* Active skin rashes or breaks in the skin at the test site.
* Active skin diseases or inflammatory skin conditions including contact dermatitis within 10cm of the test site.
* Showering or bathing after the Day -5 baseline sampling and unwilling to refrain from showering or bathing whilst at Surrey CRC (Day 0 to Day 1).
* Participation in another clinical trial within 90 days preceding randomisation.
* Pregnant or breastfeeding women.
* Any other medical condition, which in the opinion of the Investigator, should preclude participation.
* Unwillingness to fulfil the performance requirements of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Reduction of bacterial load at each test site. | 1 and 10 minutes after application.
  Reduction in bacterial load of the test product in comparison to a negative control.

SECONDARY OUTCOMES:
Persistence of reduction in bacterial load at each test site. | 30 minutes - 24 hours
  Reduction in bacterial load of the test product in comparison to a negative control over a longer duration.
Relative efficacy compared to a positive control | 1-10 minutes, and 30 minutes - 24 hours
  To assess the reduction in bacterial load after application when compared to a similar commercially available product.
Number of participants with treatment-related adverse events as assessed by a 5-point scale based on comment from the participant, and recorded assessments of erythema and oedema. | From application
  Assessed by comments from the participant logged on a five-point scale, and recorded assessments of erythema and oedema by the investigator. Erythema and oedema are each assessed on a five-point scale of none to severe.

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Bendel, Principal Investigator — Medical Director
Locations (1):
- Surrey Clinical Research Centre, Guildford, Surrey, United Kingdom